CLINICAL TRIAL: NCT06265480
Title: FallFitness Fallprevention Exercise Program for Community-dwelling Older Adults
Brief Title: FallFitness Fallprevention Program for Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dalarna University (Other)
Collaborators: Sormland County Council, Sweden (Other)
Responsible Party: Principal Investigator, Marina Arkkukangas, Researcher, Dalarna University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-04577-01
Record Dates: First submitted 2024-02-08; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Fall Injury; Fall; Self Efficacy

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Study will be singled blinded (assessors)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FallFitness intervention group (Experimental): FallFitness 8-weeks exercise program, pre-and post assessment.
  Interventions: Other: FallFitness intervention group
- Control group (No Intervention): No treatment, standard information about fall prevention, pre-and post assessment.

INTERVENTIONS:
Other: FallFitness intervention group — Eight week group-based fallprevention intervention. A total of eight session (1-hour once a week).
  Arms: FallFitness intervention group

SUMMARY:
The overall aim with this project is to collaborate with four organisations for retired persons located in a small region of middle Sweden. The project aims to test and evaluate a newly developed group-based fall prevention exercise program regarding the effects and experiences of both leading and participating in the intervention. The design of the study is a randomised controlled trial including a total of 100 participants (60+), 50 participants in the intervention and 50 participants in the control group.

DETAILED DESCRIPTION:
Research questions of interest in the project are:

1. Can an eight week (eight sessions) high intensity group based fall prevention program increase strength, balance, activity level, quality of life, self-efficacy as well as reduce sedentary behavior, fear of falling and fall frequency in older adults?
2. Can older adults learn fall techniques by participating in an eight-week (eight-session) high intensity group based fall prevention program?
3. What experiences are there from the trained leaders and the participants in the intervention?
4. How can the program be implemented in the organisations for retired persons, facilitators and barriers?

A total of at least 10 volunteers will be recruited from the organisations for retired persons and trained to be instructors of the FallFitness program. These FallFitness instructors will lead the intervention groups in the planned randomised controlled trial.

For the 50 participants randomized to the intervention group a eight program including six different central components, strength, balance, self-efficacy, motor skills, and falling technique will be introduced. Estimation of about ten participants in each group with a total of five groups are planned.

Materials needed are mainly soft judo carpets. The exercise takes place in groups and most of the exercises are done in pairs, which has been a successful concept in previously research on a similar programme, Judo4Balance.

Outcome measures of interest:

Strength, balance, quality of life, activity level, fear of falling, confidence in one's own ability to perform various activities without falling, fall frequency and falling techniques. Further a "train the trainer" approach will be evaluated for implementation and a long term perspective of fallprevention.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age
* Fluent in Swedish language in both speech and writing

Exclusion Criteria:

* Physically weak, cannot sit upright without support and/or holding up the neck in a lying position and or rolls backwards
* Coronary artery disease and unstable angina
* Recently cataract treatment

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical function by Short Physical Performance Battery | Baseline and at two months follow up
  Balance, strength and walking

SECONDARY OUTCOMES:
Self-efficacy (balance confidence) | Baseline and at two months follow up
  Falls self-efficacy
Fear of Falling | Baseline and at two months follow up
  Questionnaire
EuroQoL-5 Dimension Questionnaire (EQ-5D) | Baseline and at two months follow up
  Quality of life questionnaire
Fallfrequency | A total of 12 months falldiary from baseline
  Falldiary every month
Falling techniques | Baseline and at two months follow up
  Falling backwards and sideways
Handgrip strength | Baseline and at two months follow up
  Handgrip strength measured by hand dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Marina Arkkukangas, PhD, Principal Investigator — Dalarna University
Locations (1):
- Marina Arkkukangas, Eskilstuna, Sormland, Sweden

REFERENCES:
- [Derived] Arkkukangas M, Stromqvist Baathe K, Tonkonogi M, Liljeroos M. More Than Just Exercise: Older Adults' Experience of the Peer-Led Group-Based FallFitness Program. Clin Interv Aging. 2025 Jul 1;20:931-939. doi: 10.2147/CIA.S527142. eCollection 2025. PMID 40621091
- [Derived] Arkkukangas M, Baathe KS, Hamilton J, Hassan A, Tonkonogi M. FallFitness exercise program provided using the train-the-trainer approach for community-dwelling older adults: a randomized controlled trial. BMC Geriatr. 2024 Nov 30;24(1):983. doi: 10.1186/s12877-024-05575-0. PMID 39616365